CLINICAL TRIAL: NCT05880693
Title: Dexmedetomidine Versus Magnesium Sulfate in Controlled Hypotension During Rhinoplasty Surgeries
Brief Title: Comparisons Between Dexmedetomidine and Magnesium Sulfate in Controlled Hypotension During Rhinoplasty Surgeries
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: mohamed (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor-Investigator, mohamed, assissant professor of anesthesia, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Sameh
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Dexmedetomidine; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: 56 patients got enrolled and then divided into two groups. Group 1 received dexmedetomidine (n=28), while the group 2 received magnesium sulfate (n=28). MAP, as well as heart rate, were recorded. Surgeon satisfaction was approximated for the surgical field quality.
Who Masked: Investigator
Masking Description: 56 patients got enrolled and then divided into two groups. Group 1 received dexmedetomidine (n=28), while the group 2 received magnesium sulfate (n=28). MAP, as well as heart rate, were recorded. Surgeon satisfaction was approximated for the surgical field quality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): The first group (group 1): (n= 28): Received a loading dose of dexmedetomidine 1 μg/kg in a normal saline 0.9% solution of 100 ml 10 minutes before anesthesia induction and then a 0.4 ug/kg/h via syringe infusion pump during the time of surgery.
  .
  Interventions: Drug: Dexmedetomidine
- group 2 (Experimental): The second group (group 2): (n= 28): Received magnesium sulfate 30 mg/kg as a loading dose in a saline 0.9% solution of 100 ml infusion through the syringe pump10 minutes before anesthesia induction and then a 10 mg/kg/h via syringe infusion pump during the time of surgery
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Dexmedetomidine — Group 1 received dexmedetomidine
  Other Names: magnesium sulfate
  Arms: group 1
Drug: Magnesium sulfate — the group 2 received magnesium sulfate
  Arms: group 2

SUMMARY:
General anesthesia organizes the best option for controlled blood pressure during rhinoplasty surgery. The primary agent applied in controlling hypotension should have particular unique characteristics. The dexmedetomidine central and peripheral sympatholytic performance is usually indicated by low blood pressure and low heart rate. magnesium sulfate is among the best agents used.

DETAILED DESCRIPTION:
This is a prospective comparative randomized study. 56 patients got enrolled and then divided into two groups. Group 1 received dexmedetomidine (n=28), while the group 2 received magnesium sulfate (n=28). MAP, as well as heart rate, were recorded. Surgeon satisfaction was approximated for the surgical field quality. The amount of blood loss during the entire process was measured. The score of pain was evaluated using the NRS rating scale. Sedation score through Ramsey sedation score. The time required for the first requirement of analgesia was also recorded as well as intraoperative and postoperative problems.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old
2. ASA (American Society of Anesthesiologists) grading I and II
3. patients undergo rhinoplasty surgery under general anesthesia

Exclusion Criteria:

1. The pregnant ladies
2. patients suffering from hypertension ischemic heart diseases renal insufficiency, neuromuscular diseases, hepatic impairment
3. cerebrovascular inadequacy and diabetic neuropathy, coagulopathies,
4. patients taking antiplatelets
5. Refused study,
6. patients of age < 18 or > 60 were unauthorized from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome was to determine the bleeding score | 24 hours postoperative period
  The primary outcome was to determine the bleeding score, the secondary outcomes included the mean arterial pressure as well as heart rate aiming to arrive at a surgical field free from the blood through controlled Hypotension, determination of surgeon satisfaction, and operation time, they also aided in anesthesia recovery through the use of the Aldrete score, Ramsey sedation score, and the first analgesia postoperative requirement.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed GA aboelsuod, Principal Investigator — AZHAR
Locations (1):
- Mohamed gawad Abdel aboelsuod, Cairo, Egypt